CLINICAL TRIAL: NCT00714012
Title: Evaluation of Information Displays-A Paper, Computer and Simulator Based Study
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: Applied Medical Visualizations (Industry)
Responsible Party: Sponsor
Other Study IDs: 12002
Record Dates: First submitted 2008-07-08; First posted 2008-07-14 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-08

CONDITIONS: Healthy
Keywords: Display development; Intuitive display use; visualizations are intuitive
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1 Visualization users: End users of the domain specific visualizations.
  Interventions: Other: observational

INTERVENTIONS:
Other: observational — presented with paper-based sets, web based sets or human simulator based set of questionnaires designed to identify the users' experience level and optimal visual or auditory elements for each specific domain.

SUMMARY:
Our objective is to develop intuitive, meaningful and ergonomically efficient informative displays specific to the user's domain.

DETAILED DESCRIPTION:
Typically information monitors present numeric values, waveforms, alarms and informative sounds in a single sensor single indicator manner (5). In an effort to improve the situational awareness of the end user (6), we design and develop various visual metaphors and audible representations of information to communicate the past, present, and future status of a complex system. Our studies will identify the visual and auditory elements that optimize the presentation of critical domain specific information in an intuitive, meaningful manner as well as communicate critical events efficiently and saliently as they arise.

ELIGIBILITY:
Inclusion Criteria:

* projected end users of the domain specific visualizations.
* experts and novice users of the domain specific information.

Exclusion Criteria:

* Subjects having been exposed to a particular visualization prior to testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: projected end users of the domain specific visualizations. experts and novice users of the domain specific information.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2004-10; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Subjects will be able to identify components of the visualization from predetermined lists of answers. | At time of observation

CONTACTS AND LOCATIONS:
Overall Officials: Dwayne Westenskow, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Koch SH, Weir C, Westenskow D, Gondan M, Agutter J, Haar M, Liu D, Gorges M, Staggers N. Evaluation of the effect of information integration in displays for ICU nurses on situation awareness and task completion time: A prospective randomized controlled study. Int J Med Inform. 2013 Aug;82(8):665-75. doi: 10.1016/j.ijmedinf.2012.10.002. Epub 2013 Jan 26. PMID 23357614